CLINICAL TRIAL: NCT01180842
Title: Treatment of Anxiety/Depression and Pain Through Relaxation Yoga for Patient With CF
Brief Title: Treatment of Anxiety/Depression and Pain Through Relaxation Yoga for Patient With Cystic Fibrosis (CF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0911-104
Record Dates: First submitted 2010-05-25; First posted 2010-08-12 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Cystic Fibrosis
Keywords: CF
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alternative Treatment (Other): The CF Patient Population receiving the specific yoga study treatment
  Interventions: Other: Yoga treatment program

INTERVENTIONS:
Other: Yoga treatment program — yoga program designed specifically for the patient with CF

SUMMARY:
The investigators research question is whether or not yoga effectively alleviates symptoms of pain, sleep disturbance, anxiety and depression in children with cystic fibrosis. If yoga does prove to be effective, the investigators will educate our CF population about the benefits they may experience if they choose to incorporate yoga into their CF therapy. The investigators will also go on to do further research of other complementary alternative medicine therapies.

This is a pre/post-test study with 20 subjects. The subjects will serve as their own controls. Each subject will participate in six yoga sessions over a ten week period. Subjects' symptoms will be evaluated with the use of questionnaires. The investigators will also test cortisol levels on weeks -2, -1, 1, 6, 7, 8. Cortisol is a hormone that is affected by stress. Testing of cortisol throughout the study will help us determine the subjects' stress level throughout the study.

DETAILED DESCRIPTION:
H1: The implementation of a yoga therapy program decreases symptoms of pain within our CF population.

H2: The implementation of a yoga therapy program decreases symptoms of sleep disturbance within our CF population.

H3: The implementation of a yoga therapy program decreases symptoms of anxiety within our CF population.

H4: The implementation of a yoga therapy program decreases symptoms of depression within our CF population.

ELIGIBILITY:
Inclusion Criteria:

* Positive diagnosis of CF
* Males or females within the ages of 9 and 18

Exclusion Criteria:

* No positive diagnosis of CF
* Younger than 9 years of age or older than 18 years of age
* Concomitant illness or disease that may inhibit the patient's ability to participate in the study as determined by the principal investigator
* The patient has participated in an investigational treatment study 30 days prior to pre-session week -2.
* The patient is currently participating in yoga sessions one or more times per week.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Improve Quality of Life measured through self report questionnaires | We expect this study to last one year.
  Tool: CFQ-R

SECONDARY OUTCOMES:
Reduce symptoms of pain measured through self report questionnaires | 1 year
  Tools: 1) MSAS and 2)Additional Pain Symptoms Questions
Reduce symptoms of anxiety measured through self report questionnaires and cortisol testing | 1 year
  Assessed through 1)Saliva cortisol testing and 2)tools:STAIC and HADS
Reduce symptoms of sleep disturbance measured through self report questionnaires | 1 year
  tools: 1)MSAS and 2)CES-DC
Reduce symptoms of depression measured through self report questionnaires and cortisol testing | 1 year
  tools: 1)CES-DC, 2) HADS and 3) saliva cortisol testing

CONTACTS AND LOCATIONS:
Overall Officials: John McNamara, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota, United States